CLINICAL TRIAL: NCT06134947
Title: Assessment of Right Ventricular Function Among Children With Chronic Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khalaf Abd El Hamid Abdullah, dr, Assiut University
Other Study IDs: Right Ventricular Function in
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Right Ventricular Function
Keywords: chronic lung disease
MeSH Terms: interventions — Ventricular Function, Right

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: group A=75 patients as case group (children with Chronic Respiratory Disease)
  Interventions: Other: Echocardiographic examination
- Group B: group B=75 children as control group (children with no Chronic Respiratory Disease).
  Interventions: Other: Echocardiographic examination

INTERVENTIONS:
Other: Echocardiographic examination — Standard 2D echocardiographic evaluation of right ventricle systolic function will be performed as follows:
  * Tricuspid annular peak systolic excursion (TAPSE) will be measured by placing M- mode cursor through tricuspid annulus and measuring the amount of longitudinal motion of the annulus at the peak systole in the longitudinal apical 4chamber view, TAPSE <-2 Z Score is considered abnormal .
  * Tricuspid annular peak systolic velocity (TAPSV) by tissue Doppler <-2 Z Score is considered abnormal.
  Through Tissue Doppler Imaging values of right ventricle will be obtained from the apical four -chamber view using a sample volume placed at the lateral corner of the tricuspid annulus. Peak systolic annular velocity (Ś).
  Other Names: Echo Doppler study for right ventricular function

SUMMARY:
A Pediatric Chronic lung disease (CLD) is an abroad term that encompasses a heterogeneous group of different clinicopathological disorders that advance slowly over months or years. They can broadly be divided into two groups: those with a known cause and those without. Cystic fibrosis, broncho-pulmonary dysplasia or lung of prematurity, asthma, chronic gastro esophageal reflux/aspiration pneumonitis, and constrictive obliterative bronchiolitis, chronic infection, and hypersensitivity pneumonitis are all included in the first group. The second group is subdivided into primary pulmonary diseases (idiopathic interstitial pneumonia, persistent tachypnea of infancy associated with neuroendocrine cell hyperplasia, pulmonary lymphatic and vascular disorders, etc.) and systemic diseases with a pulmonary manifestation (e.g., Langerhans cell histio- cytosis, vasculities, and granulomatosis) Asthma is a chronic inflammatory disease of the airways which is related to airway obstruction, hyper responsiveness and characterized recurrent wheezing, coughing and breathlessness Asthma, recurrent hypoxemia, and hypercarbia, together with various mediators and cytokines released due to chronic inflammation, lead to pulmonary vasoconstriction Exaggerated respiratory efforts in asthmatic patients may increase intrathoracic pressure, which may increase right-ventricular (RV) afterload. Consequently, pulmonary hypertension may develop, which could then lead to RV hypertrophy and/or dilatation There are lacks of information's about right ventricular (RV) function in children with chronic lung diseases so in this study the RV systolic function will be evaluated. Systolic right ventricular (RV) function is an important predictor in the course of heart disease such as in pulmonary hypertension .The European Society of Cardiology and the American Society of Echocardiography recommend the use of tissue Doppler imaging for the evaluation of both diastolic and systolic functions .

DETAILED DESCRIPTION:
A Pediatric Chronic lung disease (CLD) is an abroad term that encompasses a heterogeneous group of different clinicopathological disorders that advance slowly over months or years . They can broadly be divided into two groups: those with a known cause and those without. Cystic fibrosis, bronchopulmonary dysplasia or lung of prematurity, asthma, chronic gastro esophageal reflux/aspiration pneumonitis, and constrictive obliterative bronchiolitis, chronic infection, and hypersensitivity pneumonitis are all included in the first group. The second group is subdivided into primary pulmonary diseases (idiopathic interstitial pneumonia, persistent tachypnea of infancy associated with neuroendocrine cell hyperplasia, pulmonary lymphatic and vascular disorders, etc.) and systemic diseases with a pulmonary manifestation (e.g., Langerhans cell histiocytosis, vasculitis's, and granulomatosis) .

Asthma is a chronic inflammatory disease of the airways which is related to airway obstruction, hyper responsiveness and characterized recurrent wheezing, coughing and breathlessness .

Asthma, recurrent hypoxemia, and hypercarbia, together with various mediators and cytokines released due to chronic inflammation, lead to pulmonary vasoconstriction . Exaggerated respiratory efforts in asthmatic patients may increase intrathoracic pressure, which may increase right-ventricular (RV) afterload. Consequently, pulmonary hypertension may develop, which could then lead to RV hypertrophy and/or dilatation .

Blood viscosity from polycythemia secondary to hypoxia also plays a role in the development of pulmonary hypertension.

Patients with chronic lung diseases develop pulmonary hypertension (and core-pulmonal in severe cases) because of the recurrent hypoxia and chronic inflammation this results in right heart enlargement and ventricular hypertrophy .

The initial insult in congenital diaphragmatic hernia (CDH) occurs during embryogenesis, resulting in aberrant bilateral pulmonary parenchymal and cardiovascular development, followed by ongoing inhibition of growth secondary to compression by abdominal contents. These developmental abnormalities contribute to the clinical phenotypes in CDH, with evidence of pulmonary hypoplasia, pulmonary hypertension, and ventricular dysfunction all contributing to morbidity and mortality .

According to the Cystic Fibrosis Foundation Patient Registry (CFFPR), the United States has over 30,000 people living with CF (> 70,000 worldwide) with roughly 1,000 new cases of CF diagnosed every year.

This disease primarily affects the respiratory system and the gastrointestinal system. However, recent studies suggest a direct or indirect involvement of the cardiovascular system. The destruction of lung parenchyma and pulmonary vasoconstriction due to chronic hypoxemia may result in pulmonary hypertension causing cor pulmonale. Some studies imply that the CFTR protein is also expressed in cardiac myocytes, including both atrial and ventricular myocytes .

The European Society of Cardiology and the American Society of Echocardiography recommend the use of tissue Doppler imaging for the evaluation of both diastolic and systolic functions .

However, irregular shape of the right ventricle, its retrosternal location, and the frequent coexistence of lung hyperinflation make standard "gray-scale" imaging suboptimal for routine assessment of the right ventricle .

There are lacks of information's about right ventricular (RV) function in children with chronic lung diseases so in this study the investigator will evaluate of the RV systolic function.

Systolic right ventricular (RV) function is an important predictor in the course of heart disease such as in pulmonary hypertension and RV infarction. However, one of its widely used parameters, RV ejection fraction (EF), is difficult to assess both with accuracy and ease. This is due to the complex geometrical shape of the RV.

Traditionally, RV fractional area or long-axis change measurements (FAC and FLC) by two-dimensional (2D) echocardiography have been employed, also lD parameters such as the tricuspid annular peak systolic excursion (TAPSE) . The advent of tissue Doppler imaging (TDI) has initiated long-axis function analysis of both ventricles difficult to obtain by conventional echocardiograph, whereby pulsed-wave TDI at the lateral tricuspid annulus allows the recording of RV peak myocardial contraction velocity (v)

ELIGIBILITY:
Inclusion Criteria:

* Children have aged from 7 years to 18 years.
* Patients diagnosed with chronic lung disease at pediatric pulmonology unit by chest radiograph, computerized topography (CT) chest finding, sweat chloride test and pulmonary function tests.

A total of seventy - five participants will be selected to be included at the study (group A=75 patients as case group (children with Chronic Respiratory Disease) , group B=75 children as control group (children with no Chronic Respiratory Disease).

Including:

31 patients with bronchial asthma. 22 patients with interstitial pulmonary fibrosis. 22 patients with cystic fibrosis.

Exclusion Criteria:

* Congenital heart disease and Acquired heart diseases.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sample Size Calculation:
  The sample size will be determined using epi-infoVersion 7 based on the following prerequisites:
  * Confidence level = 95%
  * Expected frequency of Chronic Respiratory Disease = 4.9%.
  * Confidence limit =5%
  * Population size = 10000.
  * Sample size (n) =75 patients as case group A total of seventy - five participants will be selected to be included at the study (group A=75 patients as case group (children with Chronic Respiratory Disease) , group B=75 children as control group (children with no Chronic Respiratory Disease).
  Including:
  31 patients with bronchial asthma. 22 patients with interstitial pulmonary fibrosis. 22 patients with cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Right ventricular function evaluation among children with chronic Lung disease | 1 year
  Right ventricular function evaluation among children with chronic Lung disease through tricuspid annular peak systolic excursion (TAPSE) and tricuspid annular peak systolic velocity (TAPSV) by tissue Doppler

REFERENCES:
- [Background] Horak F, Doberer D, Eber E, Horak E, Pohl W, Riedler J, Szepfalusi Z, Wantke F, Zacharasiewicz A, Studnicka M. Diagnosis and management of asthma - Statement on the 2015 GINA Guidelines. Wien Klin Wochenschr. 2016 Aug;128(15-16):541-54. doi: 10.1007/s00508-016-1019-4. Epub 2016 Jul 1. PMID 27370268
- [Background] Massoud TF, Hademenos GJ, De Salles AA, Solberg TD. Experimental radiosurgery simulations using a theoretical model of cerebral arteriovenous malformations. Stroke. 2000 Oct;31(10):2466-77. doi: 10.1161/01.str.31.10.2466. PMID 11022081
- [Background] Han R, Bansal D, Miyake K, Muniz VP, Weiss RM, McNeil PL, Campbell KP. Dysferlin-mediated membrane repair protects the heart from stress-induced left ventricular injury. J Clin Invest. 2007 Jul;117(7):1805-13. doi: 10.1172/JCI30848. PMID 17607357
- [Background] Nagueh SF, Appleton CP, Gillebert TC, Marino PN, Oh JK, Smiseth OA, Waggoner AD, Flachskampf FA, Pellikka PA, Evangelisa A. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. Eur J Echocardiogr. 2009 Mar;10(2):165-93. doi: 10.1093/ejechocard/jep007. No abstract available. PMID 19270053
- [Background] Patel N, Massolo AC, Kipfmueller F. Congenital diaphragmatic hernia-associated cardiac dysfunction. Semin Perinatol. 2020 Feb;44(1):151168. doi: 10.1053/j.semperi.2019.07.007. Epub 2019 Jul 30. PMID 31420110
- [Background] Warth JD, Collier ML, Hart P, Geary Y, Gelband CH, Chapman T, Horowitz B, Hume JR. CFTR chloride channels in human and simian heart. Cardiovasc Res. 1996 Apr;31(4):615-24. PMID 8689654
- [Background] Timmusk S, Paalme V, Pavlicek T, Bergquist J, Vangala A, Danilas T, Nevo E. Bacterial distribution in the rhizosphere of wild barley under contrasting microclimates. PLoS One. 2011 Mar 23;6(3):e17968. doi: 10.1371/journal.pone.0017968. PMID 21448272
- [Background] Mejza F, Gnatiuc L, Buist AS, Vollmer WM, Lamprecht B, Obaseki DO, Nastalek P, Nizankowska-Mogilnicka E, Burney PGJ; BOLD collaborators; BOLD study collaborators. Prevalence and burden of chronic bronchitis symptoms: results from the BOLD study. Eur Respir J. 2017 Nov 22;50(5):1700621. doi: 10.1183/13993003.00621-2017. Print 2017 Nov. PMID 29167298
- [Background] Koestenberger M, Ravekes W, Everett AD, Stueger HP, Heinzl B, Gamillscheg A, Cvirn G, Boysen A, Fandl A, Nagel B. Right ventricular function in infants, children and adolescents: reference values of the tricuspid annular plane systolic excursion (TAPSE) in 640 healthy patients and calculation of z score values. J Am Soc Echocardiogr. 2009 Jun;22(6):715-9. doi: 10.1016/j.echo.2009.03.026. Epub 2009 May 7. PMID 19423286